CLINICAL TRIAL: NCT05662540
Title: PET/MR in the Staging and Efficacy Evaluation of Newly Diagnosed NK/T-cell Lymphoma: a Prospective, Single-arm Clinical Study
Brief Title: PET/MR in the Staging and Efficacy Evaluation of Newly Diagnosed NK/T-cell Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NK-PETMR
Record Dates: First submitted 2022-11-13; First posted 2022-12-22 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Positron-Emission Tomography; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/MR (Experimental): This is a prospective, single-arm clinical study. Subjects who meet the inclusion criteria will receive PET/MR examination within 28 days before treatment after signing the informed consent form for pre-treatment evaluation. Stage I/II patients received PET/MR again 21-35 days after 2 and 4 courses of standard treatment for mid-term and final efficacy evaluation. Stage III/IV patients received PET/MR again 21-35 days after 3 and 6 courses of standard treatment for mid-term and final efficacy evaluation. Follow-up assessments are then continued, every 12 weeks for the first year, and every 24 weeks thereafter (clinical symptoms, physical examination, enhanced CT of the cervix, abdomen, and pelvis, and enhanced MR of the nasopharynx) until disease progression (PD), death, withdrawal of informed consent, or study finish. For subjects with suspected PD, histopathological results should be obtained whenever possible to confirm or exclude PD status.
  Interventions: Device: Positron Emission Tomography/Magnetic Resonance (PET/MR)

INTERVENTIONS:
Device: Positron Emission Tomography/Magnetic Resonance (PET/MR) — 18F-FDG PET/MR imaging (manufacturer: Siemens, model: Biography mMR). Research devices are marketed products.

SUMMARY:
This study intends to evaluate the application value of Positron Emission Tomography/Magnetic Resonance (PET/MR) in the staging and efficacy evaluation of NK/T cell lymphoma, aiming to explore a more accurate system for predicting the prognosis of patients and guiding the treatment.

DETAILED DESCRIPTION:
Nature Killer/T-cell Lymphoma (NKTCL) is a highly heterogeneous, aggressive lymphoma subtype with poor prognosis. Ninty percent of patients have lesions involving the nasal region, other extranodal organs include adrenal glands, gastrointestinal tract, skin and so on. Local tumor infiltration (bone, skin, paranasal sinus, etc) is a poor prognostic factor. Therefore, NK/T-cell lymphomas have high demands on the resolution of fine anatomical structures. PET/CT and nasopharyngeal contrast-enhanced MR are routine examination methods for diagnostic staging and efficacy evaluation, but the images cannot be fused, and the divided examinations bring inconvenience to patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed NK/T-cell lymphoma based on the WHO classification 2016
* Age from 14 to 70 years-old
* ECOG 0-2 score
* Patients with a life expectancy of at least 6 months
* Patient has not been treated before for NK/T cell lymphoma
* Commit to abide by the research procedures and cooperate with the implementation of the whole process of research
* Written informed consent

Exclusion Criteria:

- Subjects who meet any of the following criteria are not eligible for study entry

* Diagnosed aggressive NK cell leukemia
* Pregnant or lactating women
* Liver and kidney insufficiency
* Other PET/MR contraindications:

  1. Those with implanted functional electronic devices such as cardiac pacemakers
  2. Carotid aneurysm clipping and other implants are ferromagnetic materials
  3. Implanted perfusion devices such as insulin perfusion pumps
  4. Those who do not cooperate in examinations such as coma, mental illness, and critically ill patients
  5. Those who are claustrophobic
* Other concurrent and uncontrolled medical conditions that the investigator believes will affect the patient's participation in the study

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The sensitivity, specificity and accuracy of PET/MR in the staging of newly diagnosed NK/T-cell lymphoma patients | Baseline
  SUVmax, organs, et al.
The sensitivity, specificity and accuracy of PET/MR in the efficacy evaluation of newly diagnosed NK/T-cell lymphoma patients | After at least 2 cycles
  SUVmax, organs, et al.

SECONDARY OUTCOMES:
Exploratory construction of prognostic prediction or efficacy evaluation system for newly treated NK/T-cell lymphoma based on PET/MR imaging indicators. | Baseline up to data cut-off (up to approximately 4 years)
  SUVmax, organs, progression-free survival, overall survival, et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China